CLINICAL TRIAL: NCT07303179
Title: A Multicenter, Randomized Controlled Study on the Evaluation of Functional Impairment and the Promotion of Exercise Rehabilitation Standards in Maintenance Hemodialysis (MHD) Patients
Brief Title: Exercise Rehabilitation for Functional Impairment in Maintenance Hemodialysis Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Yunnan (Other)
Responsible Party: Principal Investigator, Qinyuan Deng, Resident Physician, The First People's Hospital of Yunnan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFKT-1023-005
Record Dates: First submitted 2025-09-25; First posted 2025-12-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: End-Stage Renal Disease (ESRD); Maintenance Hemodialysis (MHD)
Keywords: Exercise Rehabilitation; Maintenance Hemodialysis; Physical Function
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Rehabilitation Group (Experimental): This arm will follow the "Standards for Rehabilitation Services in CKD Patients" and receive structured exercise rehabilitation therapy (ERT) in addition to routine hemodialysis. The intervention includes three phases:
  Warm-up exercises (e.g., stretching, limb flexion/extension, leg raises),
  Core exercises (e.g., upper-limb resistance training, bedside cycling),
  Relaxation exercises (e.g., whole-body stretching).
  Each session will last 20-60 minutes, three times per week, for a total duration of two years. All sessions will be supervised by trained healthcare staff, and exercise prescriptions will be individualized according to patient condition to ensure safety and feasibility.
  Interventions: Behavioral: Exercise Rehabilitation Therapy (ERT)
- Control Group (No Intervention): Participants in this group will receive routine maintenance hemodialysis only, without any additional exercise intervention.

INTERVENTIONS:
Behavioral: Exercise Rehabilitation Therapy (ERT) — The intervention follows the "Standards for Rehabilitation Services in CKD Patients" and applies structured exercise rehabilitation therapy (ERT) in addition to routine maintenance hemodialysis. The ERT program includes three phases:
  Warm-up exercises (e.g., stretching, limb flexion/extension, leg raises),
  Core exercises (e.g., upper-limb resistance training, bedside cycling),
  Relaxation exercises (e.g., whole-body stretching).
  Each session will last 20-60 minutes, three times per week, for a total of two years.
  Other Names: Exercise Rehabilitation Therapy; Exercise Training Program
  Arms: Exercise Rehabilitation Group

SUMMARY:
Maintenance hemodialysis (MHD) is the main treatment for patients with end-stage renal disease (ESRD). Although dialysis prolongs survival, many patients experience reduced physical function, poor quality of life, and higher risks of hospitalization and death. Lack of exercise often leads to muscle weakness and disability, further burdening patients, families, and healthcare systems.

Rehabilitation medicine has shown promise in improving outcomes in patients with chronic kidney disease. Chinese experts have developed the "Standards for Rehabilitation Services in CKD Patients," which outline goals, procedures, and safety measures for exercise interventions. Based on these Standards, this study will evaluate the effects of structured exercise rehabilitation techniques (ERT) during routine dialysis.

This multicenter, randomized controlled trial will enroll 800 patients from 15 dialysis centers in China, including 40 patients at The First People's Hospital of Yunnan Province. Eligible patients will be randomly assigned to an intervention group (dialysis plus ERT) or a control group (dialysis only). ERT includes warm-up, core resistance and cycling exercises, and relaxation, performed 3 times per week for 20-60 minutes per session over 2 years.

The study will assess whether ERT can improve muscle strength, walking distance, psychological health, nutritional and cognitive status, and overall quality of life. Hospitalization and mortality will also be recorded as clinical outcomes. Results will provide scientific evidence for the feasibility, safety, and effectiveness of promoting standardized exercise rehabilitation in MHD patients.

ELIGIBILITY:
Inclusion Criteria:

1. On maintenance hemodialysis for ≥3 months.
2. Age 18-74 years.
3. Receiving adequate standard medical management.
4. Hemodialysis frequency: 3 times per week.
5. Kt/V > 1.2.

Exclusion Criteria:

1. New York Heart Association (NYHA) class IV heart failure.
2. Recent uncontrolled unstable angina.
3. Severe peripheral arterial disease or musculoskeletal disorders.
4. Walking distance <200 meters.
5. Resting oxygen saturation <90%.
6. Amputation or other conditions precluding exercise.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in 6-minute walk distance (6MWD) | From enrollment until 2 years after the end of intervention.
  Functional capacity will be assessed using the 6-minute walk test (6MWT) at baseline and every 6 months. The change in walking distance reflects improvement in functional impairment and exercise tolerance among maintenance hemodialysis (MHD) patients receiving standardized exercise rehabilitation therapy (ERT). Unit of Measure: Meters (m).
Incidence of hospitalization due to cardiovascular events | From enrollment until 2 years after the end of intervention.
  Hospitalizations caused by cardiovascular events will be recorded, including acute myocardial infarction, other acute coronary syndromes, congestive heart failure requiring hospitalization, and severe arrhythmias (e.g., complete atrioventricular block, cardiac arrest). Data will be used to assess whether ERT reduces cardiovascular morbidity. Incidence will be expressed as the proportion of participants experiencing at least one event during the follow-up period.
Incidence of cerebrovascular events | From enrollment until 2 years after the end of intervention.
  The occurrence of cerebrovascular events, including intracerebral hemorrhage, subarachnoid hemorrhage, and ischemic stroke (cardioembolic or other etiologies), will be documented and compared between the ERT and control groups. Incidence will be expressed as the proportion of participants experiencing at least one event during the follow-up period.
All-cause mortality | From enrollment until 2 years after the end of intervention.
  All-cause mortality will be monitored throughout the study to evaluate the long-term safety and prognostic impact of standardized exercise rehabilitation therapy in MHD patients. All-cause mortality will be expressed as the proportion of participants who die from any cause during the follow-up period.

SECONDARY OUTCOMES:
Change in handgrip strength | From enrollment until 2 years after the end of intervention.
  Handgrip strength will be assessed using a calibrated handgrip dynamometer. Measurements will be performed at baseline and every 6 months during the study period. The change in handgrip strength will reflect improvements in upper limb muscle strength among maintenance hemodialysis (MHD) patients receiving standardized exercise rehabilitation therapy (ERT).
  Unit of Measure: Kilograms (kg)
Change in lower limb muscle strength assessed by Five Times Sit-to-Stand Test (5STS) | From enrollment until 2 years after the end of intervention.
  Lower limb muscle strength will be assessed using the Five Times Sit-to-Stand Test (5STS). Participants will be seated on a standard armless chair (43 cm in height) with feet flat on the floor, arms crossed over the chest, and the back not supported by the chair. Upon the verbal command "start," participants will be instructed to stand up fully and sit down five times as quickly as possible. Timing will begin at the start command and stop when the participant completes the fifth stand. The time required to complete five repetitions will be recorded.
  Assessments will be performed at baseline and every 6 months during the study period. Changes in 5STS performance will reflect improvements in lower limb muscle function among maintenance hemodialysis patients receiving standardized exercise rehabilitation therapy (ERT). Unit of Measure: Seconds (s)
Change in depressive symptoms assessed by the Self-Rating Depression Scale (SDS) | From enrollment until 2 years after the end of intervention.
  Depressive symptoms will be evaluated using the Self-Rating Depression Scale (SDS), a validated self-report instrument comprising 20 items rated on a 4-point Likert scale. The total raw score is converted to a standard score, with higher scores indicating more severe depressive symptoms. Assessments will be performed at baseline and every 6 months. Changes in SDS scores will reflect the impact of exercise rehabilitation therapy (ERT) on depression among maintenance hemodialysis (MHD) patients. Unit of Measure: Score on a scale (SDS standard score range: 25-100).
Change in anxiety level assessed by the Self-Rating Anxiety Scale (SAS) | From enrollment until 2 years after the end of intervention.
  Anxiety symptoms will be assessed using the Self-Rating Anxiety Scale (SAS), a validated self-administered questionnaire consisting of 20 items. Each item is rated on a 4-point Likert scale. The total raw score is converted to a standard score, with higher scores indicating more severe anxiety symptoms. Assessments will be conducted at baseline and every 6 months during the study period. Changes in SAS scores will be used to evaluate the effect of exercise rehabilitation therapy (ERT) on anxiety levels in maintenance hemodialysis (MHD) patients. Unit of Measure: Score on a scale (SAS standard score range: 25-100).
Change in body mass index (BMI) | From enrollment until 2 years after the end of intervention.
  Body mass index (BMI) will be calculated as body weight divided by the square of height (kg/m²). Measurements will be obtained at baseline and every 6 months. Changes in BMI will be used to evaluate the impact of exercise rehabilitation therapy (ERT) on body composition and nutritional status in maintenance hemodialysis (MHD) patients. Unit of Measure: Kilograms per square meter (kg/m²).
Change in cognitive function assessed by the Montreal Cognitive Assessment (MoCA) | From enrollment until 2 years after the end of intervention.
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA) at baseline and every 6 months. The MoCA is a 30-point cognitive screening tool evaluating domains including attention, memory, language, and executive function, where higher scores indicate better cognitive performance. Changes in MoCA scores will be used to assess the effect of exercise rehabilitation therapy (ERT) on cognitive function in maintenance hemodialysis (MHD) patients. Unit of Measure: Score on a scale (MoCA score range: 0-30).
Change in self-management ability assessed by the Hemodialysis Self-Management Scale | From enrollment until 2 years after the end of intervention.
  Self-management ability will be assessed using the Hemodialysis Self-Management Scale, a 20-item patient-reported questionnaire designed to evaluate self-management behaviors in patients undergoing maintenance hemodialysis. The scale assesses domains such as treatment adherence, dietary and fluid management, symptom monitoring, and health-related behaviors. Assessments will be conducted at baseline and every 6 months during the study period. Changes in self-management scores will be used to evaluate the effect of exercise rehabilitation therapy (ERT) on self-management ability in maintenance hemodialysis (MHD) patients. Unit of Measure: Score on a scale (total score; range: 0-20)
Change in urea reduction ratio (URR) | From enrollment until 2 years after the end of intervention.
  Urea reduction ratio (URR) will be calculated based on pre- and post-dialysis blood urea levels at baseline and every 3 months to evaluate dialysis adequacy. Unit of Measure: Percent (%). Laboratory parameters are assessed every 3 months in accordance with routine clinical monitoring practices in maintenance hemodialysis patients.
Change in single-pool Kt/V for urea | From enrollment until 2 years after the end of intervention.
  Single-pool Kt/V for urea will be calculated at baseline and every 3 months using pre- and post-dialysis blood urea concentrations to assess dialysis adequacy in maintenance hemodialysis (MHD) patients receiving exercise rehabilitation therapy (ERT). Unit of Measure: Dimensionless. Laboratory parameters are assessed every 3 months in accordance with routine clinical monitoring practices in maintenance hemodialysis patients.
Change in hemoglobin concentration | From enrollment until 2 years after the end of intervention.
  Hemoglobin concentration will be measured at baseline and every 3 months to evaluate changes in anemia status in maintenance hemodialysis (MHD) patients receiving exercise rehabilitation therapy (ERT). Unit of Measure: Grams per liter (g/L). Laboratory parameters are assessed every 3 months in accordance with routine clinical monitoring practices in maintenance hemodialysis patients.
Change in serum ferritin | From enrollment until 2 years after the end of intervention.
  Serum ferritin levels will be measured at baseline and every 3 months to assess changes in iron stores in MHD patients undergoing exercise rehabilitation therapy (ERT). Unit of Measure: Nanograms per milliliter (ng/mL). Laboratory parameters are assessed every 3 months in accordance with routine clinical monitoring practices in maintenance hemodialysis patients.
Change in transferrin saturation (TSAT) | From enrollment until 2 years after the end of intervention.
  Transferrin saturation (TSAT) will be calculated at baseline and every 3 months to evaluate iron utilization in maintenance hemodialysis (MHD) patients receiving exercise rehabilitation therapy (ERT). Unit of Measure: Percent (%). Laboratory parameters are assessed every 3 months in accordance with routine clinical monitoring practices in maintenance hemodialysis patients.
Change in serum calcium | From enrollment until 2 years after the end of intervention.
  Serum calcium levels will be measured at baseline and every 3 months to assess changes in mineral metabolism in maintenance hemodialysis (MHD) patients receiving exercise rehabilitation therapy (ERT). Unit of Measure: Millimoles per liter (mmol/L). Laboratory parameters are assessed every 3 months in accordance with routine clinical monitoring practices in maintenance hemodialysis patients.
Change in serum phosphate | From enrollment until 2 years after the end of intervention.
  Serum phosphate concentrations will be measured at baseline and every 3 months to evaluate changes in mineral metabolism in maintenance hemodialysis (MHD) patients undergoing exercise rehabilitation therapy (ERT). Unit of Measure: Millimoles per liter (mmol/L). Laboratory parameters are assessed every 3 months in accordance with routine clinical monitoring practices in maintenance hemodialysis patients.
Change in intact parathyroid hormone (iPTH) | From enrollment until 2 years after the end of intervention.
  Serum intact parathyroid hormone (iPTH) levels will be measured at baseline and every 3 months to assess changes in parathyroid function and mineral bone disorder status in maintenance hemodialysis (MHD) patients receiving exercise rehabilitation therapy (ERT). Unit of Measure: Picograms per milliliter (pg/mL). Laboratory parameters are assessed every 3 months in accordance with routine clinical monitoring practices in maintenance hemodialysis patients.
Change in C-reactive protein (CRP) | From enrollment until 2 years after the end of intervention.
  Serum C-reactive protein (CRP) levels will be measured at baseline and every 3 months to assess changes in systemic inflammation associated with exercise rehabilitation therapy (ERT) in maintenance hemodialysis (MHD) patients. Unit of Measure: Milligrams per liter (mg/L). Laboratory parameters are assessed every 3 months in accordance with routine clinical monitoring practices in maintenance hemodialysis patients.
Change in serum albumin | From enrollment until 2 years after the end of intervention.
  Serum albumin concentration will be measured at baseline and every 3 months to evaluate changes in nutritional status in maintenance hemodialysis (MHD) patients receiving exercise rehabilitation therapy (ERT). Unit of Measure: Grams per liter (g/L). Laboratory parameters are assessed every 3 months in accordance with routine clinical monitoring practices in maintenance hemodialysis patients.
Change in prealbumin | From enrollment until 2 years after the end of intervention.
  Serum prealbumin levels will be assessed at baseline and every 3 months to evaluate short-term changes in nutritional status in maintenance hemodialysis (MHD) patients undergoing exercise rehabilitation therapy (ERT). Unit of Measure: Milligrams per liter (mg/L). Laboratory parameters are assessed every 3 months in accordance with routine clinical monitoring practices in maintenance hemodialysis patients.
Change in triglycerides | From enrollment until 2 years after the end of intervention.
  Serum triglyceride levels will be measured at baseline and every 3 months to assess changes in lipid metabolism in maintenance hemodialysis (MHD) patients receiving exercise rehabilitation therapy (ERT). Unit of Measure: Millimoles per liter (mmol/L). Laboratory parameters are assessed every 3 months in accordance with routine clinical monitoring practices in maintenance hemodialysis patients.
Change in total cholesterol | From enrollment until 2 years after the end of intervention.
  Total serum cholesterol levels will be measured at baseline and every 3 months to evaluate changes in lipid profile in maintenance hemodialysis (MHD) patients undergoing exercise rehabilitation therapy (ERT). Unit of Measure: Millimoles per liter (mmol/L). Laboratory parameters are assessed every 3 months in accordance with routine clinical monitoring practices in maintenance hemodialysis patients.

OTHER OUTCOMES:
Correlation between metabolomic and proteomic features and 6-minute walk distance (6MWD) | From baseline sampling to 2 years after the end of intervention.
  Untargeted metabolomic and proteomic profiling will be performed on blood samples collected at baseline and follow-up using liquid chromatography-mass spectrometry (LC-MS/MS). Normalized relative abundances of detected metabolites and proteins will be correlated with 6-minute walk distance (6MWD) measured by the 6-minute walk test. Correlation analyses will be conducted to identify molecular features associated with functional capacity and responsiveness to exercise rehabilitation therapy (ERT) in maintenance hemodialysis (MHD) patients. Unit of Measure: Correlation coefficient (Pearson or Spearman correlation will be used depending on data distribution).
Correlation between metabolomic and proteomic features and depressive symptoms (Self-Rating Depression Scale, SDS) | From baseline sampling to 2 years after the end of intervention.
  Untargeted metabolomic and proteomic profiling will be performed on blood samples collected at baseline and follow-up using LC-MS/MS. Normalized relative abundances of detected metabolites and proteins will be correlated with depressive symptom severity assessed by the Self-Rating Depression Scale (SDS). The SDS standard score ranges from 25 to 100, where higher scores indicate more severe depressive symptoms. Correlation analyses will be performed to identify molecular features associated with depressive symptoms and psychological responsiveness to ERT in MHD patients. Unit of Measure: Correlation coefficient (Pearson or Spearman correlation will be used depending on data distribution.).
Correlation between metabolomic and proteomic features and cognitive function (Montreal Cognitive Assessment, MoCA) | From baseline sampling to 2 years after the end of intervention.
  Untargeted metabolomic and proteomic profiling will be performed using LC-MS/MS. Normalized molecular feature abundances will be correlated with cognitive function assessed by the Montreal Cognitive Assessment (MoCA), a 30-point cognitive screening tool, where higher scores indicate better cognitive performance. Unit of Measure: Correlation coefficient (Pearson or Spearman correlation will be used depending on data distribution).

CONTACTS AND LOCATIONS:
Locations (1):
- The First People's Hospital of Yunnan Province, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: Clinical Research Protocol Version2 (2026-01-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT07303179/Prot_SAP_002.pdf
  • Study Protocol and Statistical Analysis Plan: Clinical Research Protocol Version1 (2025-01-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT07303179/Prot_SAP_000.pdf
  • Informed Consent Form: Revised Informed Consent Form (ICF ) Version2 (2026-01-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT07303179/ICF_003.pdf
  • Informed Consent Form: Informed Consent Form (ICF ) Version2 (2025-02-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT07303179/ICF_001.pdf